CLINICAL TRIAL: NCT06961851
Title: Feasibility Pilot of Accelerated Stimulation With TMS for Treatment of Major Depressive Disorder (FAST-MDD)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAST-MDD
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients with major depressive disorder
  Interventions: Other: aTMS utilizing the MagVenture TMS device

INTERVENTIONS:
Other: aTMS utilizing the MagVenture TMS device — Participants will complete 6 MagVenture TMS sessions per day for 5 days at the SLP Clinic. Sessions will take place with at least 30 minutes between each session. The first session will determine the baseline motor threshold for delivering aTMS. We will be stimulating the dorsolateral prefrontal cortex (DLPFC) which is within the FDA approved uses. Participants will complete a PHQ9 on all 5 treatment days and 1, 2, 4, and 6 weeks post treatment via REDCap Participants will complete daily adverse event logs via REDCap

SUMMARY:
This is a mixed-methods study that includes three steps. The first is a focus group to collect opinions and feedback about implementation of aTMS among clinicians, technicians, nurses, and other clinical staff at the St. Louis Park (SLP) clinic who are experienced with delivering TMS. The second is the delivery of a set of questionnaires delivered to TMS patients at the SLP clinic who are awaiting the start of their TMS series. The third is the delivery of aTMS utilizing the MagVenture TMS device to patients on the SLP rTMS waitlist.

The purpose of this feasibility study is to examine the acceptability and efficacy of Accelerated Transcranial Magnetic Stimulation (aTMS) delivered using an accelerated schedule. Repetitive Transcranial Magnetic Stimulation (rTMS) is traditionally delivered once a day, five days a week, for nearly 7 weeks for a total of 36 treatments. While aTMS is quick to deliver, a standard session lasting 10-20 minutes, this schedule is time intensive for patients. It often requires time off from work to accommodate daily driving time to and from the clinic as well as treatment time. This can be disruptive to a patients life and ability to attend all treatment sessions while continuing with their own life responsibilities.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Current patient of SLP Clinic
* Diagnosis of Unipolar Depression
* Have tried at least 1 antidepressant
* Ability to maintain stable medication regimen for duration of study

Exclusion Criteria:

* Has received TMS in the last 3 months
* Diagnosis of Bipolar Depression
* Any lifetime psychosis or mania
* Recent suicide attempt within 90 days of study visit
* Use of Benzodiazepines in past 4 weeks
* Presence of any contraindication to TMS assessed by the TMS Adult Safety Screen including individual history of uncontrolled seizures
* Current or history of alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
Reduction in depressive symptoms | baseline and 6 weeks
  assessed via the PHQ9, comparing baseline to end of treatment and 6 weeks post treatment.

SECONDARY OUTCOMES:
Durability data of aTMS | 0, 1, 2, 4, and 6 weeks post treatment
Dropout rate | 6 weeks
  will be calculated via completion rates

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States